CLINICAL TRIAL: NCT01705886
Title: Clinical and Economic Comparison of Robotic Versus Manual Knee Arthroplasty
Brief Title: Clinical and Economic Comparison of Robot Assisted Versus Manual Knee Replacement
Status: Completed | Type: Observational
Sponsor: Northwest Surgical Specialists, Vancouver (Other)
Collaborators: Stryker Surgical Corp (Unknown)
Responsible Party: Sponsor
Other Study IDs: MAKO-02; 2015-004 (Other: Stryker)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Knee Arthroplasty
Keywords: Osteoarthritis; Joint Disease; Arthritis; Musculoskeletal Disease; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Arthritis; Musculoskeletal Diseases; Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee Arthroplasty: Patients undergoing knee replacement surgery. This may be a Total Knee Arthroplasty or MAKO® Robot Assisted Medial Knee Arthroplasty.
  The MAKO® Robot Assisted surgeries use the RESTORIS Multicompartmental Knee System.
  The total knee arthroplasty uses the Depuy Knee Replacement System or the Stryker® Knee Replacement System.
  Interventions: Procedure: Total Knee Arthroplasty; Procedure: MAKO® Robot Assisted Medial Knee Arthroplasty; Device: RESTORIS Multicompartmental Knee System; Device: Depuy Knee Replacement System; Device: Stryker® Knee Replacement System

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Patients undergoing manual (no robot used) surgery to replace of all 3 compartments of the knee
  Other Names: TKA; Total Knee Replacement
Procedure: MAKO® Robot Assisted Medial Knee Arthroplasty — Patients undergoing a MAKO® robot assisted surgery to replace the medial compartment of the knee
  Other Names: unilateral knee arthroplasty (UKA)
Device: RESTORIS Multicompartmental Knee System — The RESTORIS Multicompartmental Knee (MCK) System components are intended for single or multicompartmental knee replacement used in conjunction with the MAKO® Robotic Arm Interactive Orthopedic System (RIO®). The components can be used for medial compartment, lateral compartment, patellofemoral compartment, or bicompartmental (medial and patellofemoral compartments) knee replacement. The device is intended to be used with bone cement.
  Other Names: RESTORIS® MCK MultiCompartmental Knee System; FDA 501K number K090763
Device: Depuy Knee Replacement System — The Depuy Knee Replacement System components are intended for use in total knee replacement. These components are intended for implantation with bone cement.
Device: Stryker® Knee Replacement System — The Stryker® Knee Replacement System components are intended for use in total knee replacement. These components are intended for implantation with bone cement.

SUMMARY:
The purpose of this study is to document and compare the surgical and after surgery costs, recovery time, and outcomes of two procedure types:

* Robotic assisted surgery replacing one compartment of the knee
* Manual (robot is not used) surgery replacing all three compartments of the knee (total knee replacement)

The hypothesis is that robot assisted partial knee replacement is cost effective and provides clinical outcomes that are equivalent to a manual total knee replacement.

DETAILED DESCRIPTION:
Background and Significance:

The primary indications for joint replacement surgery include severe lower extremity pain that prevents individuals from performing normal daily activities. The level of pain experienced by these patients cannot be managed successfully with oral medications, physical therapy, or joint injections of steroids or hyaluronic acid. The source of the pain most commonly is a result of arthritic changes in the joint; the arthritis may be due to osteoarthritis, rheumatoid arthritis, or traumatic arthritis. Patients who are appropriate candidates for partial joint replacement surgery also may experience joint stiffness that interferes with their normal daily activities. In addition, there usually is radiographic evidence of changes in the joint caused by the arthritic process. Joint damage is evaluated radiographically in order to classify the severity of the joint disease. Partial joint replacement surgery is performed to replace the diseased parts of the joint with prosthesis. There are a variety of options that surgeons and patients can choose for their joint replacement surgery. There are many different joint replacement component systems manufactured by several different companies; some systems are recommended for particular types of patients while others can be used in a greater number of patients. Recently, new techniques have been introduced that are classified as minimally invasive because they require smaller surgical incisions to implant standard joint prostheses. Patients who are younger, thinner, and in better overall health are usually the best surgical candidates for minimally invasive procedures.

Osteoarthritis affects 40 million Americans and 15 million people in the United States suffer from degenerative arthritis of the knee. Unicondylar knee arthroplasty (UKA) was introduced as a treatment option for degenerative arthritis of the knee in the early 1970's[1]. The procedure initially yielded variable results and this unpredictability resulted in broadly low levels of usage[1]. Recent improvements in the surgical techniques and technology used for UKA have increased the effectiveness of this surgery. As the average age of the United States population increases, this surgical procedure will become even more common. It is estimated by the Millennium Research Group that there will be 55,100 unicondylar knee procedures in 2010 and the compound annual growth rate from 2009 to 2014 will be 8.3%.

UKA knee arthroplasty can be viewed as an attractive alternative to total knee arthroplasty (TKA) assuming the patient's osteoarthritis has remained isolated in a single compartment or two compartments. UKA knee arthroplasty are generally less invasive procedures than TKA. Since the procedure is less invasive there is usually less blood loss; more cartilage, tissue, and bone is sparred, which results in shorter recovery times than TKA. This procedure is attractive to adults who are interested in remaining active pain-free lifestyles as they age.

The cost-effectiveness of healthcare interventions, especially new technology, is becoming essential. Comparing the procedural costs of robotic-assisted surgery and the outcomes of the patients versus TKA, the gold standard, will help substantiate whether robotic-assisted surgery from an economic viewpoint is a cost-effective treatment. In addition the rehabilitation after knee replacement surgery is critical to achieving proper functional outcomes. Information pertaining to knee replacement post discharge costs has been limited. Due to the lack of studies and the continued growth in the number of knee arthroplasty surgeries it is imperative to track post discharge costs of all variables. We will be documenting and comparing the procedural and postoperative costs, recovery time, and outcomes of three procedure types in robotic assisted unicompartmental knee arthroplasty, robotic assisted bicompartmental knee arthroplasty and manual total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age, 21-80 years
* Sex, males and females will be included
* BMI less than or equal to 39
* Stable health, the patient would be able to undergo surgery and participate in the follow-up program based on physical examination and medical history
* Patient is willing and able to cooperate in follow-up therapy at Rebound facilities in Vancouver, WA
* Patient has stable and functional collateral ligaments
* Patient or patient's legal representative has signed the Informed Consent form
* Failed non-operative management of their joint disease
* Need to obtain pain relief and improved function
* Moderate or severe pain with either walking or at rest
* Diagnosed with osteoarthritis in one or more compartments of the knee and non-surgical treatment options have failed to provide relief for symptoms
* Patient exhibits preoperative radiographic evidence of joint degeneration that cannot be treated in non-operative fashion

Exclusion Criteria:

* Patients who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in the study
* Patients with pre-op flexion contracture greater than 10 degrees, overall flexion less than 115 degrees, and varus/valgus greater than 10 degrees
* Patient who is on workmen's compensation
* Patients who are on chronic long acting preoperative narcotic pain medication
* Patients with inflammatory polyarthritis
* Women who are pregnant
* Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes
* Subjects who are currently involved in another clinical study with the exception to an outcomes study
* Patients with a pathology which, in the opinion of the Principal Investigator, will adversely affect healing
* A diagnosed systemic disease that would affect their welfare or the overall outcome of study (i.e. Paget's disease, renal osteodystrophy)
* Patients receiving an isolated patellofemoral UKA,lateral UKA, or bi-compartmental arthroplasty
* Patients with significant medical condition preventing a well-functioning contralateral knee
* cognitively unable to complete study health-related quality of life forms

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and non-pregnant females undergoing knee replacement who are between 21 and 80 years of age with stable health and are willing and able to have physical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-10; Primary Completion 2018-01 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Cost per case at 1 year | 1 year
  Cost per case for 1 year. The inpatient costs, analgesic use, physical therapy, durable medical equipment, and postoperative visits will be used to calculate the cost at 1 year.

SECONDARY OUTCOMES:
American Knee Society Knee Score | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year after surgery
  The American Knee Society Score is an assessment and questionnaire that provides a rating of the pain, function, range of motion, and knee joint stability. It is subdivided into a knee score that rates only the knee joint itself and a functional score that rates the patient's ability to walk and climb stairs.

OTHER OUTCOMES:
Reduced WOMAC | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year after surgery
  The Reduced WOMAC is a truncated version of the Western Ontario and McMaster's University Osteoarthritis Index. The questionnaire is designed to assess pain, disability and joint stiffness in the osteoarthritis patient.
Knee injury and Osteoarthritis Outcome Score | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year after surgery
  The KOOS or Knee injury and Osteoarthritis Outcome Score are patient completed questionnaires which assess the patient's opinion regarding their knee and its associated osteoarthritis.
EQ-5D | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year after surgery
  The EQ-5D is a standardized instrument for use as a measure of health outcome.
Forgotten Joint Score | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year after surgery
  The Forgotten Joint Score is a 12-item questionnaire completed by the patient to determine how aware they are of their joint in their everyday life.
Length of Stay | At inpatient discharge which has an expected average of 2 days after surgery
  Number of days patient stayed in hospital after surgery
Time to physical therapy discharge | At discharge from physical therapy which has an expected average of 6 weeks after surgery
  Days after surgery to meet physical therapy discharge criteria of
  * Range of motion 5 to 115 degrees
  * Strength 4/5 for flexion and extension expressed as a percent of maximal isometric contraction from pre-operative assessment and determined with a dynamometer
  * Gait with minimal limp without an assistive device for a distance of 250 feet
  * Able to ascend/ descend a flight of stairs with step over gait with good control (and with use of handrail)
Timed Up and Go | 1-2 weeks prior to surgery, 6 weeks after surgery, 3 months after surgery
  Timed up and Go (TUG) Test: Participants are instructed to stand up from a seated position from a standard chair, walk 3 m around a cone and then return to the chair and resume a seated position. Pace is self-selected. The time to complete the test is recorded.
6 Minute Walk Test (6MWT) | 1-2 weeks prior to surgery, 6 weeks after surgery, 3 months after surgery
  Participants are instructed to cover as much distance walking in 6 minutes and can stop and rest if necessary. The course is 30 meters in length, marked at 1 meter intervals with cones marking the turn around point. Distance measured is rounded up to the nearest meter and recorded.
Stair Ascend/Descend Test | 1-2 weeks prior to surgery, 6 weeks after surgery, 3 months after surgery
  Participants are asked to ascend and descend 11 steps using a hand rail if necessary. Stair height is 17.8 cm (7"). Pace is self selected. The time to ascend/ descend 1 flight of stairs is recorded.
Return to Driving Time | 6 weeks after surgery
  Number of days from surgery until patient returned to driving. In addition if the knee replacement procedure was a performed on the left leg or right leg will be documented because this could factor into time it takes to return to driving.
Return to Work Time | 6 weeks after surgery
  The number of days from surgery to return to work.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Borus, MD, Principal Investigator — Northwest Surgical Specialists / Rebound Orthopedics and Neurosurgery; Donald Roberts, MD, Principal Investigator — Northwest Surgical Specialists / Rebound Orthopedics and Neurosurgery
Locations (1):
- Rebound Orthopedics and Neurosurgery, Vancouver, Washington, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT01705886/Prot_SAP_000.pdf
  • Informed Consent Form (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT01705886/ICF_001.pdf